CLINICAL TRIAL: NCT06786052
Title: Efficacy of Probiotics on Postprandial Energy Metabolism of Adults With Overweight or Obesity: an EXploratory Clinical Trial
Brief Title: EXploratory Study on Postprandial Energy Metabolism
Acronym: EXPEM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: Centre de recherche en nutrition humaine de Rhône-Alpes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: L-029
Record Dates: First submitted 2025-01-08; First posted 2025-01-22 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Obesity and Overweight; Moderately Obese
Keywords: Metabolic health; Probiotics; Postprandial metabolism
MeSH Terms: conditions — Obesity; Overweight | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): The product contains the probiotic strain and no other ingredients.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): The control product is a placebo with the same characteristics of appearance and packaging as the tested product.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — After randomization, participants will consume the probiotic for 3 months.
  Arms: Probiotic
Dietary Supplement: Placebo — After randomization, participants will consume the placebo for 3 months.
  Arms: Placebo

SUMMARY:
This exploratory, double-blinded clinical trial on 66 randomized adults aged 50 to 70 years with moderate overweight or obesity but considered metabolically healthy will consist of comparing metabolic and microbiota parameters before and after 3 months of consumption of a probiotic or a placebo.

DETAILED DESCRIPTION:
This study will focus on adults (men and postmenopausal women) aged 50 to 70 years who are overweight or moderately obese (BMI between 27 and 34.9 kg/m2) and considered metabolically healthy.

66 participants will be recruited according to the following inclusion and exclusion criteria. There will be a total of 5 visits and the study participation will last about 3.5 months.

The main hypothesis is that daily supplementation of the probiotics for 3 months in the defined population will improve certain parameters related to the cardiometabolic profile such as glucose tolerance and lipemia during the postprandial phase, compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Man or woman;
2. Age between 50 and 70 years old (inclusively);
3. Postmenopausal women, i.e. with amenorrhea for more than a year with no identified cause
4. BMI between 27 and 34.9 kg/m2 (inclusively);
5. Stable weight in the last 3 months (+/- 5% of total body weight);
6. Waist circumference ≥ 80 cm for women, ≥ 94 cm for men;
7. Sedentary to moderately active (less than 30 minutes of moderate physical activity, 3 times a week);
8. Agreeing not to consume fermented or supplemented foods (including bifidus yogurts and other foods supplemented with probiotics), dietary supplements (high in fiber (prebiotics), high protein, or other food supplements that may interact with the gut microbiota or energy metabolism), laxatives and any substance that can control metabolic parameters such as weight, blood glucose or lipid metabolism during the study period (from the screening visit);
9. Agreeing to receive probiotics or placebo supplementation randomly;
10. Able to understand the information given, read and write in French and have signed the informed consent form;
11. Agreeing to submit to the entire study protocol;
12. Having fibre consumption (through diet or supplementation) of less than 30g/day;
13. Having a freezer to store stool samples before the visit.

Exclusion Criteria:

1. Participant with unstable medical or psychological conditions that, in the opinion of the investigator, could lead the participant to be non-compliant or uncooperative during the study or that could compromise the safety or participation in the study (according to articles L.1121-6, L.1121-8, L.1121-9 and L1122-1-2 of the Public Health Code);
2. Presence of pathology detectable on clinical examination and medical questioning that may interfere with the study endpoints;
3. Alcohol consumption exceeding 30g of alcohol/day (1 dose of alcoholic beverage = 10g of alcohol) or abuse or dependence on another proven drug;
4. Tobacco consumption (or vaping equivalent) > to 5 cigarettes per day and inability to restrict smoking or vaping on the exploratory days provided for in the protocol;
5. Failure to comply with the exclusion period for another study specified in the "national volunteer file";
6. Adult subject to a legal protection measure (guardianship, curatorship);
7. Person deprived of liberty by a judicial or administrative decision;
8. Person who has exceeded the annual amount of compensation in the year for participation in research protocols;
9. Person not affiliated to a social security system or beneficiary of a similar system;
10. Absence of valid approved health proof(s) in the event of government measures in an exceptional epidemic situation;
11. Person with a specific diet (vegetarian, lacto-vegetarian, vegan, high-protein, etc.);
12. People consuming food supplements (pre or probiotics, or minerals (divalent cations such as magnesium and calcium)) regularly during the month prior to the screening visit;
13. Blood donation within 2 months prior to the screening visit;
14. Claustrophobic to the point that indirect calorimetry measurement cannot be done;
15. Person with limited venous access that can make it difficult to draw blood and insert a catheter;
16. Type 1 or 2 diabetes;
17. Systolic blood pressure≥ 140 mmHg;
18. Diastolic blood pressure≥ 90 mmHg;
19. Treatment for hypertension or dyslipidemia;
20. Known endocrine pathology that may interfere with carbohydrate metabolism (uncontrolled dysthyroidism, acromegaly, hypercorticism, etc.);
21. People with gastrointestinal pathologies with an inflammatory component or associated with malabsorption;
22. People suffering from bloody diarrhoea;
23. Exocrine pancreatic insufficiency;
24. People who have had intestinal or abdominal surgery (apart from appendectomy and simple hernias), bariatric surgery (gastric banding, calibrated vertical gastroplasty and sleeve gastrectomy accepted if done more than 5 years ago);
25. Severe eating disorders (e.g., anorexia/bulimia, uncontrolled binge eating syndrome, noctophagia);
26. Chronic kidney failure;
27. Hepatocellular insufficiency;
28. Immunocompromised individuals (e.g., those with AIDS, lymphoma, patients on long-term corticosteroid therapy, patients undergoing chemotherapy and allogeneic transplants);
29. Patients with central venous catheters and post-surgical patients;
30. Hematological, gastrointestinal, hepatic, neurological, or psychiatric clinically significant according to the investigator;
31. Drug treatments for obesity in the last 3 months or prescribed for the duration of the study;
32. Taking antibiotics in the month preceding the explorations (for the so-called common antibiotics of the beta-lactam family) or in the 3 months preceding the explorations according to the investigator's judgment (for other families of antibiotics);
33. Taking antidepressants in the 2 months prior to the explorations or prescribed for the duration of the study;
34. Daily intake of laxatives in the 3 months prior to explorations or other medications that may strongly interfere with the composition of the gut microbiota;
35. Taking a treatment that may interfere with the study measures, according to the judgment of the co-investigating physicians of the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in postprandial triglyceridemia after 3 months | 12 weeks
  The difference (delta) from baseline in the area under the incremental curve (AUCi (0-300 min)) of postprandial triglyceridemia in response to a test meal after 12 weeks of probiotic supplementation versus placebo.

SECONDARY OUTCOMES:
Change in vital parameter | 12 weeks
  Changes in pulse measured at baseline and at the end of intervention, with additional measurements at 1-month and 2-month intervals to monitor progress.
Change in vital parameter | 12 weeks
  Change in blood pressure measured at baseline and at the end of intervention, with additional measurements at 1-month and 2-month intervals to monitor progress.
Change in anthropometric measurement | 12 weeks
  BMI calculated in kg/m^2 by measuring the weight and height at baseline and at the end of intervention, with additional measurements at 1-month and 2-month intervals to monitor progress.
Change in anthropometric measurement | 12 weeks
  Waist-to-hip ratio calculated by measuring the waist and hip circumference at baseline and at the end of intervention, with additional measurements at 1-month and 2-month intervals to monitor progress.
Change in blood lipid concentrations from baseline | 12 weeks
  Blood samples will be collected at each visit to report lipid concentrations such as plasma/serum triglycerides, total cholesterol, HDL cholesterol, LDL cholesterol and non-esterified fatty acids.
Change in blood metabolic parameters from baseline | 12 weeks
  Blood samples will be collected at each visit to report metabolic parameters such as glucose, insulin, Hba1c and ApoB.
Change in body composition | 12 weeks
  Changes in body composition at baseline and at the end of intervention, with additional measurements at 1-month and 2-month intervals to monitor progress. It is measured using multifrequency bio-impedancemetry which quantifies the total body water and the percentages of lean and fat mass.
Change in inflammatory parameters | 12 weeks
  Changes in the plasma concentrations of TNF-α, IL6, and CRP measured at baseline and at the end of intervention, with additional measurements at 1-month and 2-month intervals for CRP.
Change in intestinal barrier integrity biomarker | 12 weeks
  Change in the plasma concentration of Zonuline measured at baseline and at the end of intervention.
Change in safety plasma concentration | 12 weeks
  Blood samples will be taken each visit in order to report safety plasma concentration, which includes the measurements of creatinine, GFR, urea, AST, ALT, gamma GT, bilirubin, albumin, and PAL.
Change in fasting exhaled gases | 12 weeks
  Changes in the levels of CO2, H2, and CH4 measured at baseline and at the end of intervention.
Change in complete blood count | 12 weeks
  Changes in the complete blood count measured throughout the intervention period.
Change in gut microbiota | 12 weeks
  Collected stool samples will be used for microbiota analysis, which allows to assess changes in the composition and diversity of the gut microbiota throughout the intervention period, as well as probiotic strain detection.
Change in postprandial kinetics of metabolic parameters | 12 weeks
  Changes in the maximum and minimum values during the postprandial period for the following parameters: glucose (time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 min), insulin (time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 min), and total cholesterol (time t0, 30, 60, 120, 180, 240, 300 min).
Change in postprandial kinetics of metabolic parameters | 12 weeks
  Changes in the peak or nadir times during the postprandial period for the following parameters: glucose (time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 min), insulin (time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 min), and total cholesterol (time t0, 30, 60, 120, 180, 240, 300 min).
Change in postprandial kinetics of metabolic parameters | 12 weeks
  Changes in the total and incremental AUCs 0-120 min, 120-300 min, and 0-300 min during the postprandial period for the following parameters: glucose (time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 min), insulin (time t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 min), and total cholesterol (time t0, 30, 60, 120, 180, 240, 300 min).
Change in postprandial kinetics of metabolic parameters | 12 weeks
  Changes in kinetics of the following parameters measured at specific time points: glucose (t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 min), insulin (t-30, 0, 15, 30, 45, 60, 90, 120, 180, 240, 300 min), and total cholesterol (t0, 30, 60, 120, 180, 240, 300 min).
Change in postprandial triglyceride levels and kinetics | 12 weeks
  Change in the maximum and minimum values as well as times at peak or nadir, total AUC 0-120 min, 120-300 min, 0-300 min during the postprandial period and triglyceride kinetics (time t-30, 0, 30, 60, 120, 180, 240, 300 min).
Change in plasma metabolome | 12 weeks
  Change in the plasma metabolome (about 1000 metabolites from 39 different classes) measured throughout the intervention period.
Assessment of average daily food intake | 12 weeks
  Assessing the average daily food intake of macronutrients and micronutrients using 3-day dietary surveys of the week prior to a visit.
Change in resting energy metabolism | 12 weeks
  Change in resting energy metabolism measured by indirect calorimetry at baseline and at the end of intervention.
Assessment of digestive tolerance | 12 weeks
  Evaluation of digestive tolerance via Gastrointestinal Symptom Assessment Scale throughout the intervention period.
Evaluation of changes in stool assessment | 12 weeks
  Evaluation of the change in stool consistency and frequency reported via Bristol and Likert scale throughout the intervention period.
Physical Activity Assessment | 12 weeks
  Physical activity assessed throughout the intervention period using International Physical Activity Questionnaire (IPAQ).
Evaluation of eating behaviour | 12 weeks
  Eating behaviour and satietogenic effect will be assessed throughout the intervention period using Three-Factor Eating Questionnaire (TFEQ-R21) and Food Cravings Questionnaires (FCQ-T and FCQ-S).
Assessment of general well-being | 12 weeks
  General well-being assessed throughout the intervention period using 36-Item Short Form Health Survey (SF-36) questionnaire.
Assessment of stress level | 12 weeks
  General stress level assessed throughout the intervention period using Perceived Stress Scale (PSS) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhône-Alpes (CRNH-RA), Pierre-Bénite, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No